CLINICAL TRIAL: NCT03189121
Title: Effect of Isocaloric Ultra Processed Versus Unprocessed Diets on Insulin Sensitivity
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170107; 17-DK-0107
Record Dates: First submitted 2017-06-15; First posted 2017-06-16 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Obesity
Keywords: Metabolism; Macronutrients; Obesity; Energy Expenditure; Glucose
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: 20 overweight and obese adult men

SUMMARY:
Background:

Increases in obesity, diabetes, and some metabolic disorders may be linked to how much processed foods people eat. Researchers want to learn more about how processed foods affect metabolic health.

Objective:

To learn about how a processed versus unprocessed diet affects the body.

Eligibility:

Men ages 18-50 with stable weight and risk factors for diabetes

Design:

Participants will be screened over 3 visits. Screening includes:

* Medical history and physical exam
* Heart and blood tests
* Psychiatric questions
* Questions about eating, sleeping, and economic status
* Riding a stationary bike
* Trying a sample meal

Between screenings, participants will eat prepared meals. They will wear an accelerometer to measure physical activity. They will write down what foods they eat and monitor their weight.

Participants will have two 4-week stays in the clinic. They will:

* Eat a special diet
* Have activity and weight monitored
* Drink water and collect urine samples to measure how many calories they are burning
* Have resting energy expenditure measured with a clear hood over the head
* Have a scan to measure body fat and bone density using low-dose x-rays
* Have a scan on a table that slides into a metal cylinder in a strong magnetic field. They will get earplugs for the loud noises.
* Have an ultrasound test to measure blood vessels
* Have insulin and glucose infused into an arm vein. Blood will be taken over 10 hours through a plastic tube in the wrist. This will happen 4 times.
* Spend multiple 24-hour periods in a room that measures oxygen used and carbon dioxide produced.
* Give blood, urine and stool samples
* Answer questionnaires and do computer tasks

DETAILED DESCRIPTION:
Nutrition science is beginning to place less emphasis on the nutrient composition of the diet and more emphasis on its comprising foods. A particular public health concern involves the consumption of foods that result from extensive industrial processing. Ultra-processed foods have become increasingly common and now contribute the majority of calories consumed in America. The rise in the prevalence of obesity, type 2 diabetes, and metabolic syndrome over the past several decades is believed to have been caused, in part, by the parallel increase in production, advertising, and consumption of ultra-processed foods. However, the metabolic effects of industrial processing per se, independent of diet calories or macronutrient composition, have not been carefully investigated in a controlled feeding study. Therefore, we will conduct an inpatient controlled feeding study in 20 overweight and obese adult men to investigate the changes in multi-organ insulin sensitivity and hepatic triglyceride content resulting from consuming two test diets for a pair of 3 week periods. The test diets will be implemented in a randomized, crossover design with each test diet following a 1 week run-in period of inpatient controlled feeding of a standard metabolic diet. The test diets will be matched for calories, macronutrient composition, sugar, fiber, and sodium, but one diet will be composed of ultra-processed foods whereas the other diet will be unprocessed foods. Multi-organ insulin sensitivity and hepatic triglyceride content will be measured at the end of each 1 week run-in period as well as at the end of each 3 week test diet period.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adult men, age 18-50 years
  2. Weight stable (< plus or minus 5 % over past 6 months)
  3. Body mass index (BMI) greater than or equal to 25 kg/m^2
  4. Plasma triglycerides > 150 mg/dl (Caucasian) or >140 mg/dl (African American)
  5. Homeostatic model of insulin resistance (HOMA-IR) > 2
  6. Able to complete daily bouts of stationary cycling at a moderate rate and intensity with a HR equal to or greater than 0.3x(220-age-HRrest)+HRrest but not exceeding 0.6x(220-age- HRrest)+HRrest and no signs of arrhythmia
  7. Written informed consent
  8. Willing to eat all the food provided in the study
  9. Willing to cease their habitual caffeine intake during the study, beginning one week prior to each inpatient admission

EXCLUSION CRITERIA:

1. Evidence of metabolic or cardiovascular disease, or disease that may influence metabolism (e.g. cancer, diabetes, thyroid disease)
2. Body weight >400 lbs. (weight limit of magnetic resonance spectroscopy gantry)
3. Taking any prescription medication or other drug that may influence metabolism (e.g. diet/weight-loss medication, asthma medication, blood pressure medication, psychiatric medications, corticosteroids, or other medications at the discretion of the PI and/or study team)
4. Hematocrit < 40%
5. Participating in a regular exercise program (> 2h/week of vigorous activity)
6. Caffeine consumption > 300 mg/day
7. Regular use of alcohol (> 2 drinks per day), tobacco (smoking or chewing) amphetamines, cocaine, heroin, or marijuana over past 6 months
8. Past or present history of eating disorder (including binge eating) or psychiatric disease, including claustrophobia since part of the protocol will involve being confined to a small room for whole-body indirect calorimetry and being in an MRI scanner for liver fat measures
9. Implants, devices, or foreign objects implanted in the body that interfere with the Magnetic Resonance procedures.
10. Volunteers with strict dietary concerns (e.g. vegetarian or kosher diet, food allergies)
11. Volunteers unwilling or unable to give informed consent
12. Non-English speakers due to unavailability of required questionnaires in other languages.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20 overweight and obese adult men.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
To determine changes in hepatic insulin sensitivity following a 3-week ultra-processed diet as compared to following 3 weeks of an unprocessed diet matched for calories, macronutrient composition, sugar, fiber, and sodium. | ongoing

SECONDARY OUTCOMES:
To determine changes in hepatic triglyceride content following a 3-week ultra-processed diet as compared to 3 weeks of an unprocessed diet matched for calories, macronutrient composition, sugar, fiber, and sodium | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hall, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Monteiro CA, Moubarac JC, Cannon G, Ng SW, Popkin B. Ultra-processed products are becoming dominant in the global food system. Obes Rev. 2013 Nov;14 Suppl 2:21-8. doi: 10.1111/obr.12107. PMID 24102801
- [Background] Tavares LF, Fonseca SC, Garcia Rosa ML, Yokoo EM. Relationship between ultra-processed foods and metabolic syndrome in adolescents from a Brazilian Family Doctor Program. Public Health Nutr. 2012 Jan;15(1):82-7. doi: 10.1017/S1368980011001571. Epub 2011 Jul 14. PMID 21752314